CLINICAL TRIAL: NCT05766293
Title: Application of Extracorporeal Shockwaves on Human Gingival Fibroblasts in Vitro Study
Brief Title: ESWT on Human Gingival Fibroblasts
Acronym: ESWT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Prabhuji MLV (Other)
Responsible Party: Sponsor-Investigator, Dr Prabhuji MLV, Professor, Head of Periodontology, Principle investigator, Clinical Professor, Krishnadevaraya College of Dental Sciences & Hospital
Organization: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: KCDS/48
Record Dates: First submitted 2023-02-14; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Periodontal Attachment Loss
Keywords: Cell culture; ESWT; Cell proliferation; Cell viability
MeSH Terms: conditions — Periodontal Attachment Loss; Hyperplasia

STUDY DESIGN:
Intervention Model Description: PCS-201-018 Fibroblast cell line (n=10) would be exposed to shockwave generator depending on Test group. Control group Fibroblast cell line (n=10) would be assessed without shockwave exposure. Cell proliferation and Cell viability will be assessed for both Test and Control Fibroblast cell lines using Scratch assay, MTT analysis and ATP analysis, accordingly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave treated group (Active Comparator): Effect of Extracorporeal shockwaves on Fibroblast cell proliferation and cell viability
  Interventions: Device: extracorporeal shockwave device
- No shockwave group (Placebo Comparator): Fibroblast cell lines assessed for proliferative rate and viability without shockwave exposure.
  Interventions: Other: Fibroblast cell lines not subjected to shockwaves from extracorporeal shockwave device

INTERVENTIONS:
Device: extracorporeal shockwave device — Fibroblast cell lines (n=10) were subjected to Shockwaves from extracorporeal shockwave device
  Arms: Shockwave treated group
Other: Fibroblast cell lines not subjected to shockwaves from extracorporeal shockwave device — Fibroblast cell lines (n=10) without shockwave exposure
  Arms: No shockwave group

SUMMARY:
The idea of treating different deformities or diseases in the maxillofacial region with Extracorporeal Shockwave Therapy (ESWT) has recently become popular. Shockwave therapy was first introduced in Germany in 1980s and has been widely used in medical practice for the management of urolithiasis, cholelithiasis and in head and neck region for sialolithiasis.

The present study 'Application of Extracorporeal Shock Wave Therapy on human gingival derived fibroblasts In-vitro study' was done to explore and evaluate the effect of shockwaves. Further, these cells were assessed for Cell - Cell interaction and Cell Viability.

In this in-vitro study, 20 fibroblast cells were included. 10 samples were considered for Control group and the remaining 10 samples were considered as Test group. Extracorporeal shockwave was applied to the Test samples. They were further analysed

DETAILED DESCRIPTION:
BACKGROUND:

Improved understanding of human biology at the molecular level, scientific and technologic advances are emerging aspects in dentistry. The idea of treating different deformities or diseases in the maxillofacial region with Extracorporeal Shockwave Therapy (ESWT) has recently become popular. Shockwave therapy was first introduced in Germany in 1980s and has been widely used in medical practice for the management of urolithiasis, cholelithiasis and in head and neck region for sialolithiasis.

AIM:

The present study 'Application of Extracorporeal Shock Wave Therapy on human gingival tissue derived fibroblasts In-vitro study' was done to explore and evaluate the effect of shockwaves. Further, fibroblast cells were assessed for Cell - Cell interaction and Cell Viability.

MATERIALS AND METHODS:

In this in-vitro study, 20 fibroblast cells were included. 10 samples were considered for Control group and the remaining 10 samples were considered as Test group. Extracorporeal shockwave was applied to the Test samples. They were further analysed using wound scratch assay which was used to assess Cell proliferative rate and scratch closure through live imaging. MTT assay and ATP assay was used to determine Cell viability after exposure to shockwaves.

ELIGIBILITY:
Inclusion Criteria:

* Viable human gingival fibroblast
* Healthy gingival tissue

Exclusion Criteria:

* contaminated samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Fibroblast cell lines exposed to shockwave from extracorporeal shockwave device | 74 hrs
  Cell proliferation and Cell viability

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya College of Dental Science and Hospital, Bengaluru, Karnataka, India